CLINICAL TRIAL: NCT00283842
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel-Group, 13-Week, Adaptive-Design Study of 4 Fixed Oral Doses of DVS SR in Adult Outpatients With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained-release (DVS SR) in Adult Outpatients With Pain Associated With Diabetic Peripheral Neuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: business reasons
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3151A5-322
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Diabetic Neuropathies; Pain
Keywords: neuropathic pain; diabetic peripheral neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- desvenlafaxine succinate sustained-release (DVS SR) 50mg (Experimental)
  Interventions: Drug: DVS SR
- desvenlafaxine succinate sustained-release (DVS SR) 100mg (Experimental)
  Interventions: Drug: DVS SR
- desvenlafaxine succinate sustained-release (DVS SR) 200mg (Experimental)
  Interventions: Drug: DVS SR
- desvenlafaxine succinate sustained-release (DVS SR) 400mg (Experimental)
  Interventions: Drug: DVS SR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DVS SR
  Arms: desvenlafaxine succinate sustained-release (DVS SR) 100mg; desvenlafaxine succinate sustained-release (DVS SR) 200mg; desvenlafaxine succinate sustained-release (DVS SR) 400mg; desvenlafaxine succinate sustained-release (DVS SR) 50mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of DVS SR in the treatment of neuropathic pain associated with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 or 2
* Painful symptoms of diabetic neuropathy in the lower extremities extremities for at least 6 months

Exclusion Criteria:

* Major Depression
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (50):
- United States (50):
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Encino, California
  - Newport Beach, California
  - Walnut Creek, California
  - Pueblo, Colorado
  - New Britain, Connecticut
  - Stratford, Connecticut
  - Waterbury, Connecticut
  - Fort Myers, Florida
  - Palm Beach Gardens, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Lawrenceville, Georgia
  - Roswell, Georgia
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - Des Moines, Iowa
  - Madisonville, Kentucky
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Albany, New York
  - Flushing, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Collegeville, Pennsylvania
  - Feasterville, Pennsylvania
  - Harleysville, Pennsylvania
  - Warwick, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Midvale, Utah
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Lakewood, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Allen R, Sharma U, Barlas S. Clinical experience with desvenlafaxine in treatment of pain associated with diabetic peripheral neuropathy. J Pain Res. 2014 Jun 23;7:339-51. doi: 10.2147/JPR.S55682. eCollection 2014. PMID 25018648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited January 2006 to February 2008
Pre-assignment Details: Participants were screened during a 7- to 28-day period, a treatment period.
Groups:
- Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg: 50mg tablets of desvenlafaxine succinate sustained-release (DVS SR) taken orally
- Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg: 100mg tablets of desvenlafaxine succinate sustained-release (DVS SR) taken orally
- Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg: 200mg tablets of desvenlafaxine succinate sustained-release (DVS SR) taken orally
- Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg: 400mg tablets of desvenlafaxine succinate sustained-release (DVS SR) taken orally
Period: Overall Study
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo
Started | 63 | 87 | 99 | 69 | 90
Completed | 51 | 69 | 68 | 42 | 75
Not Completed | 12 | 18 | 31 | 27 | 15
Not completed — Adverse Event | 8 | 7 | 21 | 21 | 5
Not completed — Protocol Violation | 1 | 5 | 4 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 5 | 4
Not completed — Lack of Efficacy | 1 | 3 | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 2 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo | Total
Number analyzed (Participants) | 63 | 87 | 99 | 69 | 90 | 408
Age Continuous [Mean (Standard Deviation); unit: years] | 61.62 (8.59) | 60.66 (9.23) | 59.80 (9.38) | 61.14 (10.03) | 58.98 (8.51) | 60.31 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 30 | 17 | 25 | 108
  Male | 47 | 67 | 69 | 52 | 65 | 300

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Pain Severity Score From Baseline to 13 Weeks
Description: Pain severity measured on a Numeric Rating Scale (NRS). Range: 0 (no pain) to 10 (worst possible pain). Change: score at 13 weeks minus score at baseline.
Time Frame: Baseline and 13 weeks
Population: The analysis population was the intent to treat.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo
Number analyzed (Participants) | 49 | 65 | 70 | 40 | 72
units on scale | -2.41 (0.26) | -2.42 (0.23) | -2.93 (0.22) | -2.74 (0.27) | -1.83 (0.22)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 50mg; Test type: Superiority or Other; p = 0.084, Hochberg
Statistical Analysis 2: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 100mg; Test type: Superiority or Other; p = 0.084, Hochberg
Statistical Analysis 3: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 200mg; Test type: Superiority or Other; p = 0.001, Hochberg
Statistical Analysis 4: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 400mg; Test type: Superiority or Other; p = 0.027, Hochberg

2. Secondary Outcome: Number of Patients With ≥50% Reduction in Mean Pain Severity Score.
Description: Pain severity measured on a Numeric Rating Scale (NRS). Range: 0 (no pain) to 10 (worst possible pain). Assessment of reduction based on change in score at 13 weeks compared to baseline.
Time Frame: Baseline and 13 weeks
Population: The analysis population is the intent to treat.
Measure: Number; unit: patients
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo
Number analyzed (Participants) | 63 | 86 | 99 | 68 | 89
patients | 22 | 32 | 36 | 22 | 23
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 50mg; Test type: Superiority or Other; p = 0.375, Hochberg
Statistical Analysis 2: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 100mg; Test type: Superiority or Other; p = 0.342, Hochberg
Statistical Analysis 3: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 200mg; Test type: Superiority or Other; p = 0.342, Hochberg
Statistical Analysis 4: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg vs Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg; Statistical analysis provided for 400mg; Test type: Superiority or Other; p = 0.375, Hochberg

ADVERSE EVENTS:
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 1 | 3 | 6
Other Adverse Events (participants affected / at risk) | 47 | 65 | 82 | 63 | 68
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo
Angina pectoris (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Ventricular tachycardia (Cardiac disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Pneumonia (Infections and infestations) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Ankle fracture (Injury, poisoning and procedural complications) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Overdose (Injury, poisoning and procedural complications) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Stress fracture (Injury, poisoning and procedural complications) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Blood glucose increased (Investigations) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Mental status changes (Psychiatric disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Urinary retention (Renal and urinary disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Orthostatic hypotension (Vascular disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Desvenlafaxine Succinate Sustained-release (DVS SR) 50mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 100mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 200mg | Desvenlafaxine Succinate Sustained-release (DVS SR) 400mg | Placebo
Abdominal pain (General disorders) | 3/63 | 2/87 | 1/99 | 1/69 | 1/90
Abscess (General disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Accidental injury (General disorders) | 3/63 | 5/87 | 7/99 | 8/69 | 6/90
Allergic reaction (General disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Asthenia (General disorders) | 4/63 | 8/87 | 9/99 | 10/69 | 4/90
Back pain (General disorders) | 2/63 | 0/87 | 3/99 | 1/69 | 5/90
Cellulitis (General disorders) | 1/63 | 1/87 | 0/99 | 0/69 | 0/90
Chest pain (General disorders) | 0/63 | 2/87 | 0/99 | 0/69 | 1/90
Chills (General disorders) | 1/63 | 0/87 | 3/99 | 0/69 | 0/90
Cyst (General disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Face edema (General disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 1/90
Fever (General disorders) | 0/63 | 1/87 | 1/99 | 1/69 | 0/90
Flu syndrome (General disorders) | 1/63 | 3/87 | 1/99 | 0/69 | 0/90
Generalized edema (General disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Headache (General disorders) | 5/63 | 7/87 | 9/99 | 5/69 | 9/90
Infection (General disorders) | 3/63 | 7/87 | 7/99 | 3/69 | 1/90
Malaise (General disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Medication error (General disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Mucous membrane disorder (General disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Neck pain (General disorders) | 0/63 | 1/87 | 0/99 | 2/69 | 0/90
Neoplasm (General disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 2/90
Overdose (General disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Pain (General disorders) | 5/63 | 3/87 | 4/99 | 3/69 | 2/90
Photosensitivity reaction (General disorders) | 0/63 | 0/87 | 0/99 | 2/69 | 0/90
Withdrawal syndrome (General disorders) | 0/63 | 0/87 | 1/99 | 1/69 | 0/90
Angina pectoris (Cardiac disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 1/90
Arrhythmia (Cardiac disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Atrial flutter (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
AV block first degree (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Bundle branck block (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Cardiovascular physical finding (Cardiac disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Coronary artery disorder (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Electrocardiogram abnormal (Cardiac disorders) | 1/63 | 0/87 | 2/99 | 0/69 | 0/90
Hemorrhage (Vascular disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Hypertension (Vascular disorders) | 2/63 | 6/87 | 11/99 | 9/69 | 7/90
Hypotension (Vascular disorders) | 1/63 | 0/87 | 0/99 | 1/69 | 1/90
Palpitation (Cardiac disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 1/90
Peripheral vascular disorder (Vascular disorders) | 1/63 | 0/87 | 2/99 | 2/69 | 0/90
Postural hypotension (Vascular disorders) | 1/63 | 2/87 | 5/99 | 4/69 | 1/90
QRS prolongation (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
QT interval prolonged (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 2/90
Sinus bradycardia (Cardiac disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Syncope (Cardiac disorders) | 0/63 | 0/87 | 1/99 | 1/69 | 0/90
Tachycardia (Cardiac disorders) | 1/63 | 1/87 | 0/99 | 5/69 | 0/90
Vasodilatation (Vascular disorders) | 1/63 | 1/87 | 4/99 | 2/69 | 0/90
Ventricular extrasystoles (Cardiac disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Ventricular tachycardia (Cardiac disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Abdominal distension (Gastrointestinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 1/90
Anorexia (Gastrointestinal disorders) | 2/63 | 3/87 | 5/99 | 3/69 | 2/90
Colitis (Gastrointestinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Constipation (Gastrointestinal disorders) | 3/63 | 4/87 | 6/99 | 6/69 | 0/90
Diarrhea (Gastrointestinal disorders) | 5/63 | 6/87 | 7/99 | 6/69 | 9/90
Dry mouth (Gastrointestinal disorders) | 2/63 | 4/87 | 5/99 | 9/69 | 2/90
Dyspepsia (Gastrointestinal disorders) | 1/63 | 3/87 | 3/99 | 1/69 | 3/90
Dysphagia (Gastrointestinal disorders) | 0/63 | 0/87 | 1/99 | 1/69 | 0/90
Eructation (Gastrointestinal disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 2/90
Flatulence (Gastrointestinal disorders) | 2/63 | 2/87 | 0/99 | 0/69 | 0/90
Gastroenteritis (Gastrointestinal disorders) | 1/63 | 1/87 | 2/99 | 2/69 | 1/90
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Gastrointestinal carcinoma (Gastrointestinal disorders) | 1/63 | 0/87 | 1/99 | 0/69 | 0/90
Gastrointestinal disorder (Gastrointestinal disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Hiatal hernia (Gastrointestinal disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Increased appetite (Gastrointestinal disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Nausea (Gastrointestinal disorders) | 9/63 | 11/87 | 27/99 | 12/69 | 2/90
Periodontal abscess (Gastrointestinal disorders) | 0/63 | 2/87 | 0/99 | 0/69 | 1/90
Retching (Gastrointestinal disorders) | 0/63 | 1/87 | 0/99 | 1/69 | 0/90
Tenesmus (Gastrointestinal disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Tooth disorder (Gastrointestinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Vomiting (Gastrointestinal disorders) | 3/63 | 3/87 | 10/99 | 2/69 | 2/90
Thyroid carcinoma (Endocrine disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Thyroid disorder (Endocrine disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Anemia (Blood and lymphatic system disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Ecchymosis (Blood and lymphatic system disorders) | 0/63 | 0/87 | 1/99 | 1/69 | 0/90
Leukopenia (Blood and lymphatic system disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Lymphadenopathy (Blood and lymphatic system disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Creatinine increased (Metabolism and nutrition disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Gout (Metabolism and nutrition disorders) | 0/63 | 1/87 | 0/99 | 1/69 | 1/90
Healing abnormal (Metabolism and nutrition disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Hypercholesteremia (Metabolism and nutrition disorders) | 2/63 | 3/87 | 3/99 | 0/69 | 1/90
Hyperglycemia (Metabolism and nutrition disorders) | 2/63 | 1/87 | 1/99 | 0/69 | 2/90
Hyperkalemia (Metabolism and nutrition disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Hyperlipemia (Metabolism and nutrition disorders) | 4/63 | 6/87 | 7/99 | 5/69 | 8/90
Hyperuricemia (Metabolism and nutrition disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Hypoglycemia (Metabolism and nutrition disorders) | 1/63 | 0/87 | 0/99 | 3/69 | 0/90
Hypokalemia (Metabolism and nutrition disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Hyponatremia (Metabolism and nutrition disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Peripheral edema (Metabolism and nutrition disorders) | 2/63 | 2/87 | 0/99 | 0/69 | 2/90
Weight gain (Metabolism and nutrition disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Weight loss (Metabolism and nutrition disorders) | 0/63 | 0/87 | 1/99 | 4/69 | 0/90
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/63 | 2/87 | 2/99 | 2/69 | 6/90
Arthritis (Musculoskeletal and connective tissue disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Joint disorder (Musculoskeletal and connective tissue disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Leg cramps (Musculoskeletal and connective tissue disorders) | 4/63 | 3/87 | 3/99 | 2/69 | 2/90
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1/63 | 0/87 | 0/99 | 2/69 | 1/90
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/63 | 1/87 | 1/99 | 0/69 | 1/90
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Myalgia (Musculoskeletal and connective tissue disorders) | 1/63 | 2/87 | 1/99 | 1/69 | 1/90
Myasthenia (Musculoskeletal and connective tissue disorders) | 1/63 | 0/87 | 1/99 | 0/69 | 0/90
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Abnormal dreams (Nervous system disorders) | 1/63 | 2/87 | 3/99 | 1/69 | 0/90
Anxiety (Nervous system disorders) | 3/63 | 0/87 | 3/99 | 0/69 | 1/90
Apathy (Nervous system disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Ataxia (Nervous system disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Carpal tunnel syndrome (Nervous system disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Confusion (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Depersonalization (Nervous system disorders) | 0/63 | 0/87 | 2/99 | 0/69 | 0/90
Depression (Nervous system disorders) | 0/63 | 2/87 | 0/99 | 1/69 | 1/90
Dizziness (Nervous system disorders) | 1/63 | 7/87 | 18/99 | 18/69 | 9/90
Emotional liability (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 3/90
Euphoria (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Hostility (Nervous system disorders) | 2/63 | 0/87 | 1/99 | 0/69 | 0/90
Hyperkinesia (Nervous system disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Hypertonia (Nervous system disorders) | 1/63 | 0/87 | 0/99 | 1/69 | 0/90
Hypesthesia (Nervous system disorders) | 0/63 | 1/87 | 3/99 | 0/69 | 2/90
Incoordination (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Insomnia (Nervous system disorders) | 3/63 | 1/87 | 4/99 | 7/69 | 1/90
Libido decreased (Nervous system disorders) | 0/63 | 1/87 | 3/99 | 1/69 | 0/90
Memory impairment (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Mental status changes (Nervous system disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Motion sickness (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Movement disorder (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Nervousness (Nervous system disorders) | 1/63 | 1/87 | 3/99 | 2/69 | 0/90
Neuralgia (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Paresthesia (Nervous system disorders) | 0/63 | 0/87 | 2/99 | 0/69 | 0/90
Reflexes decreased (Nervous system disorders) | 2/63 | 0/87 | 0/99 | 2/69 | 2/90
Reflexes increased (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Restless legs syndrome (Nervous system disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 1/90
Somnolence (Nervous system disorders) | 3/63 | 9/87 | 9/99 | 7/69 | 2/90
Thinking abnormal (Nervous system disorders) | 0/63 | 0/87 | 1/99 | 2/69 | 0/90
Tremor (Nervous system disorders) | 1/63 | 0/87 | 2/99 | 1/69 | 0/90
Twitching (Nervous system disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Vertigo (Nervous system disorders) | 1/63 | 2/87 | 2/99 | 0/69 | 0/90
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1/63 | 0/87 | 0/99 | 3/69 | 0/90
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1/63 | 4/87 | 1/99 | 2/69 | 6/90
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/63 | 2/87 | 1/99 | 0/69 | 1/90
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/63 | 1/87 | 1/99 | 0/69 | 0/90
Nose dryness (Respiratory, thoracic and mediastinal disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0/63 | 0/87 | 2/99 | 1/69 | 3/90
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Pulmonary physical finding (Respiratory, thoracic and mediastinal disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0/63 | 2/87 | 3/99 | 1/69 | 1/90
Sinusittis (Respiratory, thoracic and mediastinal disorders) | 0/63 | 3/87 | 4/99 | 1/69 | 1/90
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2/63 | 3/87 | 2/99 | 1/69 | 7/90
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Yawn (Respiratory, thoracic and mediastinal disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Acne (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 3/90
Alopecia (Skin and subcutaneous tissue disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Dry skin (Skin and subcutaneous tissue disorders) | 0/63 | 1/87 | 0/99 | 1/69 | 0/90
Eczema (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Folliculitis (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Fungal dermatitis (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 2/69 | 0/90
Furunculosis (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Herpes simplex (Skin and subcutaneous tissue disorders) | 2/63 | 0/87 | 0/99 | 0/69 | 1/90
Herpes zoster (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Nail disorder (Skin and subcutaneous tissue disorders) | 0/63 | 1/87 | 0/99 | 1/69 | 0/90
Night sweats (Skin and subcutaneous tissue disorders) | 1/63 | 1/87 | 1/99 | 0/69 | 0/90
Pruritus (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 3/99 | 3/69 | 2/90
Rash (Skin and subcutaneous tissue disorders) | 1/63 | 0/87 | 0/99 | 4/69 | 3/90
Seborrhea (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Skin benign neoplasm (Skin and subcutaneous tissue disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Skin discoloration (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Skin disorder (Skin and subcutaneous tissue disorders) | 2/63 | 0/87 | 2/99 | 0/69 | 0/90
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 2/90
Sweating (Skin and subcutaneous tissue disorders) | 3/63 | 2/87 | 7/99 | 5/69 | 1/90
Urticaria (Skin and subcutaneous tissue disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Vesiculobullous rash (Skin and subcutaneous tissue disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Abnormal vision (Eye disorders) | 0/63 | 1/87 | 1/99 | 2/69 | 0/90
Conjunctivitis (Eye disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Ear disorder (Ear and labyrinth disorders) | 1/63 | 0/87 | 1/99 | 1/69 | 0/90
Ear pain (Ear and labyrinth disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Eye pain (Eye disorders) | 0/63 | 0/87 | 0/99 | 0/69 | 1/90
Mydriasis (Eye disorders) | 0/63 | 0/87 | 0/99 | 2/69 | 0/90
Otitis media (Ear and labyrinth disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Refraction disorder (Eye disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Retinal disorder (Eye disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Taste perversion (Ear and labyrinth disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Tinnitus (Ear and labyrinth disorders) | 1/63 | 0/87 | 1/99 | 3/69 | 0/90
Abnormal ejaculation/orgasm (Reproductive system and breast disorders) | 0/63 | 0/87 | 2/99 | 1/69 | 0/90
Anorgasmia (Reproductive system and breast disorders) | 0/63 | 1/87 | 2/99 | 1/69 | 0/90
Breast disorder (Reproductive system and breast disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Cervix disorder (Reproductive system and breast disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Creatine clearance decreased (Renal and urinary disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Cystitis (Renal and urinary disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Dysuria (Renal and urinary disorders) | 1/63 | 1/87 | 2/99 | 0/69 | 0/90
Hematuria (Renal and urinary disorders) | 3/63 | 0/87 | 1/99 | 1/69 | 1/90
Impotence (Renal and urinary disorders) | 1/63 | 4/87 | 2/99 | 3/69 | 1/90
Kidney function abnormal (Renal and urinary disorders) | 0/63 | 0/87 | 1/99 | 1/69 | 0/90
Nocturia (Renal and urinary disorders) | 0/63 | 1/87 | 1/99 | 1/69 | 0/90
Prostatic disorder (Reproductive system and breast disorders) | 0/63 | 3/87 | 2/99 | 4/69 | 1/90
Prostatic specific antigen increase (Reproductive system and breast disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Pyuria (Renal and urinary disorders) | 1/63 | 0/87 | 0/99 | 0/69 | 0/90
Sexual function abnormal (Reproductive system and breast disorders) | 0/63 | 2/87 | 1/99 | 1/69 | 0/90
Testis disorder (Reproductive system and breast disorders) | 0/63 | 0/87 | 1/99 | 0/69 | 0/90
Urinary frequency (Renal and urinary disorders) | 2/63 | 0/87 | 2/99 | 1/69 | 1/90
Urinary hesitation (Renal and urinary disorders) | 0/63 | 1/87 | 1/99 | 2/69 | 0/90
Urinary incontinence (Renal and urinary disorders) | 0/63 | 1/87 | 1/99 | 1/69 | 0/90
Urinary retention (Renal and urinary disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Urinary tract infection (Renal and urinary disorders) | 1/63 | 2/87 | 1/99 | 0/69 | 3/90
Urination impaired (Renal and urinary disorders) | 0/63 | 0/87 | 1/99 | 3/69 | 0/90
Urine abnormality (Renal and urinary disorders) | 1/63 | 0/87 | 1/99 | 0/69 | 0/90
Vulvovaginal disorder (Reproductive system and breast disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Allergic reaction other than drug (General disorders) | 0/63 | 0/87 | 0/99 | 1/69 | 0/90
Local reaction to procedure (General disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 1/90
Positive event (General disorders) | 0/63 | 1/87 | 0/99 | 0/69 | 0/90
Albuminuria (Renal and urinary disorders) | 1/63 | 0/87 | 0/99 | 1/69 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication